CLINICAL TRIAL: NCT05998512
Title: Integrating Molecular, Genomic, Morphology and Environmental Features to Improve Precision Diagnosis and Treatment in Interstitial Lung Diseases (PRECISION-ILD)
Acronym: PRECISION-ILD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Responsible Party: Principal Investigator, Maria Molina, Head of Interstitial Lung Diseases Unit, Institut d'Investigació Biomèdica de Bellvitge
Other Study IDs: PMP/00083
Record Dates: First submitted 2023-07-21; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Interstitial Lung Disease; Interstitial Fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational register — This is a non-interventional observational registry on patients

SUMMARY:
Integrating Molecular, Genomic, Morphology and Environmental Features to Improve Precision Diagnosis and Treatment in Interstitial Lung Diseases (PRECISION-ILD)

Background: Interstitial Lung Diseases (ILDs) are a heterogeneous group of >100 different, rare diseases, which share the fate of progressive scarring and, ultimately, death. Two anti-fibrotic drugs have demonstrated to slow-down fibrotic progression and steroids/immunosuppressants are commonly used for inflammatory-driven ILDs. However, patient's response to therapeutic options is variable and unpredictable. Similarly, setting a correct diagnosis is difficult in most cases, especially when patients are too sick for invasive procedures.

Objectives: (1) To investigate the differences and commonalities in genetic, genomic and environmental exposures/lifestyle in fibrotic ILDs depending on the entity, disease behavior (progressive fibrosis) and treatment response; (2) To integrate the biomarkers that most impact on prognosis and treatment response in diagnostic algorithms; and (3) To explore the feasibility and cost of implementing a P4 strategy in clinical practice for fibrotic ILDs.

Methods: The investigators will extend, update and unify existing ILD cohorts (Spanish SEPAR ILD Reg, Observatory IPF.cat, CIBERES IPF and Familial ILD cohorts) in whom the researchers will: (1) record demographic, epidemiological, clinical, physiological and lung morphology (radiological +/- histological) information; (2) obtain genetic variation, telomere length, and serum protein markers; (3) investigate environmental exposures (including air-pollution), (4) apply to integrative analytical methods to identify endotypes, predictive biomarkers of disease trajectories, theragnostic biomarkers and new therapeutic targets. Results (5) will be validated in other fibrotic ILD cohorts (e.g.EuILDRegistry, Mexican fibrotic ILD Registry). Besides, the investigators will explore how to translate this P4 medicine approach in clinical practice; (6) implementing a predictive score for prognosis and improving the diagnostic approach through biological data to reduce invasive procedures, and (7) estimate educational requirement and potential health cost implications.

Viability:This project is viable because: (1) cohorts already exist and can be expanded and updated; (2) investigators have ample expertise in translational research and actively participate in ILD consortia; (3) required knowledge and methodology is already in being used by the consortium.

Clinical relevance: Due to the lethality, high social and economic burden of fibrotic ILDs, identifying the best diagnostic and therapeutic approach through preventive, personalized and precise measures is a unique opportunity to improve survival in these patients and efficiency of health-care resources.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years
* Signed informed consent
* Diagnosis of fibrotic ILD of any type in the 12 months prior to inclusion.
* Radiologic fibrotic changes of at least 5% on chest CT scan
* Ability to comply with the study protocol (in the opinion of the investigator)
* Ability to understand the information given and to sign the informed consent form.

Exclusion Criteria

* Severe, advanced stage or life-limiting chronic diseases prior to the diagnosis of fibrotic ILD, or that represent a high risk of death in the short term (one year after inclusion), such as could be metastatic oncological metastatic diseases, advanced dementia, neurodegenerative diseases in a limiting phase.
* Pregnancy or breastfeeding
* Inability to complete required visits.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients older than 18 years with diagnosis of fibrotic ILD of any type in the 12 months prior to inclusion, and radiologic fibrotic changes of at least 5% on chest CT scan.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences and commonalities in genetic, genomic and environmental exposures/lifestyle in fibrotic ILDs depending on the entity, disease behavior (progressive fibrosis) and treatment response | 3 years
  Record demographic, epidemiological, clinical, physiological and lung morphology (radiological +/- histological) information. Obtain genetic variation, telomere length, and serum protein markers. Investigate environmental exposures (including air-pollution)
Integration of the biomarkers that most impact on prognosis and treatment response in diagnostic algorithms | 3 years
  Integrative analytical methods to identify endotypes, predictive biomarkers of disease trajectories, theragnostic biomarkers and new therapeutic targets.
Feasibility and cost of implementing a P4 strategy in clinical practice for fibrotic ILDs | 3 years
  Development of a predictive score for prognosis and improving the diagnostic approach through biological data to reduce invasive procedures, and estimation educational requirement and potential health cost implications.

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital La Princesa, Madrid
  - Hospital Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No